CLINICAL TRIAL: NCT05257993
Title: An Open-label, Dose-finding, Phase Ib Study to Assess the Safety, Tolerability of JPI-547, a Dual Inhibitor of PARP/Tankyrase, in Combination With Modified FOLFIRINOX (mFOLFIRINOX) or Gemcitabine-nab-paclitaxel (GemAbraxne) in Patients With Locally Advanced and Metastatic Pancreatic Cancer
Brief Title: Study to Assess the Safety, Tolerability of JPI-547 in Combination With Modified FOLFIRINOX or Gemcitabine-nab-paclitaxel in Patients With Locally Advanced and Metastatic Pancreatic Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Onconic Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JPI-547-102
Record Dates: First submitted 2022-02-03; First posted 2022-02-25 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Pancreatic Ductal Adenocarcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (mFOLFIRINOX) (Experimental): JPI-547 and Combination Chemotherapy(mFOLFIRINOX) The study is conducted in a 3+3 dose escalation method.
  Interventions: Drug: JPI-547; Drug: modified FOLFIRINOX
- Arm B (GemAbraxane) (Experimental): JPI-547 and Combination Chemotherapy (Gemcitabine-nab-paclitaxel) The study is conducted in a 3+3 dose escalation method.
  Interventions: Drug: JPI-547; Drug: Gemcitabine-nab-paclitaxel

INTERVENTIONS:
Drug: JPI-547 — * Subjects are administered this investigational product once a week for 5 days, and have wash-out period for 2 days (5 Days on-2 Days off).
  * The investigational product is administered orally in a fasting state for 2 hours before and after meals at the same time (e.g., a certain time in the morning).
  * Capsules should be swallowed whole and should not be chewed, crushed or split.
Drug: modified FOLFIRINOX — * After IV administration of Oxaliplatin 65 mg/m2 for 2 hours
  * After IV administration of Leucovorin 400 mg/m2 for 2 hours + IV administration of Irinotecan 135 mg/m2 for 90 minutes (Irinotecan is started 30 minutes after the start of Leucovorin administration and administered simultaneously during the last 90 minutes of Leucovorin administration, but administered separately using a Y-connector without mixing)
  * Continuous IV infusion of 5-FU 2400 mg/m2 for 46 hours
  * Repeated administration every 2 weeks on a 14-day cycle
  Arms: Arm A (mFOLFIRINOX)
Drug: Gemcitabine-nab-paclitaxel — * After IV administration of nab-paclitaxel 125 mg/m2 for 30 minutes
  * IV administration of Gemcitabine 1000 mg/m2 for 30 minutes
  * Administration on Days 1, 8, and 15 on a 28-day cycle
  Arms: Arm B (GemAbraxane)

SUMMARY:
The purpose of this study is to assess the safety, tolerability of JPI-547 in combination with modified FOLFIRINOX (mFOLFIRINOX) or Gemcitabine-nab-paclitaxel (GemAbraxne) in patients with locally advanced and metastatic pancreatic cancer

DETAILED DESCRIPTION:
In combination with JPI-547 and chemotherapy in patients with locally advanced/metastatic pancreatic cancer,

Primary Objectives

* To determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D).
* To select the optimal combination chemotherapy based on the safety profile.

Secondary Objectives

* To assess the safety and toxicity.
* To evaluate anti-tumor activity.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed inoperable locally advanced or metastatic pancreatic ductal adenocarcinoma (PDAC)
2. Those with at least one measurable lesion in accordance with RECIST 1.1
3. Those with Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
4. Those with an expected survival period ≥12 weeks
5. Patients with adequate hematologic function, renal and hepatic function confirmed by the following criteria (During the screening period, laboratory tests can be retested only once.)
6. Those who voluntarily decide to participate in this clinical study after hearing sufficient explanations and who consent in writing

Exclusion Criteria:

1. Those with a history of severe hypersensitivity to the investigational product or combination anticancer drugs.
2. Those with the following medical history or surgical history/procedural history confirmed

   1. Other primary malignant tumors other than pancreatic cancer
   2. Major surgery that requires general anesthesia or breathing aid
   3. Severe cardiovascular disease
   4. New York Heart Association Class 3 or 4 heart failure
   5. Severe cerebrovascular disease t
   6. Pulmonary thrombosis, deep vein thrombosis, or bronchial asthma, obstructive pulmonary disease, and other life-threatening severe lung diseases
   7. Infections requiring administration of systemic antibiotics or antivirals, etc.
   8. Hematologic malignancy
3. Those with the following diseases

   1. Massive ascites, pleural effusions requiring therapeutic paracentesis
   2. Neuropathy ≥Grade 2
   3. Diarrhea, chronic inflammatory bowel disease
   4. Intestinal paralysis, intestinal obstruction
   5. Diseases that make oral administration difficult or affect absorption
   6. Interstitial lung disease, pulmonary fibrosis
   7. Dialysis patient
   8. Patients with clinically significant symptoms or uncontrolled central nervous system or brain metastases

   j. Uncontrolled hypertension (systolic blood pressure > 150 mmHg or diastolic blood pressure >90 mmHg) k. Bleeding diatheses l. Active hepatitis B or C virus. m. Known human immunodeficiency virus (HIV) positive
4. Those with a medication history of the following drugs

   1. Anti-cancer drug therapy such as chemotherapy and biological therapy
   2. Radiation therapy within 2 weeks of baseline
   3. Those who are taking or expected to require administration of strong inhibitors or inducers of CYP3A4
   4. (For mFOLFIRINOX cohort) Those who are taking or expected to require administration of sorivudine
   5. Patients who require continuous administration of non-steroidal anti-inflammatory drugs (NSAIDs) with high bleeding risk
   6. Patients requiring continuous administration of systemic corticosteroid equivalent to prednisone >10 mg/day
   7. Those who have received antithrombotic agents, including antiplatelet agents, anticoagulants, etc.
5. Pregnant women, lactating women, or women of childbearing potential and men who do not intend to practice abstinence or use appropriate contraceptive methods for until 6 months for men and 9 months for women after administration of the investigational product and during the clinical study
6. Those who have administered other investigational products or have received investigational medical device procedures within 4 weeks of the baseline
7. Other patients who are inappropriate or unable to participate in this clinical study at the discretion of the investigator

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-30 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D). | From the date of administration to 4 weeks (DLT period)
  The MTD is determined according to the traditional 3+3 rule-based method for each combination therapy, and it is defined as the highest dose with a DLT incidence of less than 1/3 or 2/6 subjects.

SECONDARY OUTCOMES:
To assess the adverse events, drug adverse events, and serious adverse events evaluated by NCI-CTCAE v5.0 | Until 4 weeks after the last dose administration
To evaluate anti-tumor activity. | Evaluation at 8 weeks intervals through study completion from the date of study entry until the date of progression, up to 18 months
  Anti-tumor activity is evaluated according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

CONTACTS AND LOCATIONS:
Locations (4):
- South Korea (4):
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Samsung Medical Center, Seoul
  - Seoul national university hospital, Seoul
  - Severance Hospital, Seoul